CLINICAL TRIAL: NCT06256393
Title: Cohorte Nantaise de Maladies Inflammatoires Chroniques Intestinales
Brief Title: Inflammatory Bowel Disease Cohort in Nantes
Acronym: CELESTE
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0467
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease; Ulcerative colitis; Cohort; Biocollection pathophysiology
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients of both sexes, over 18 years of age, with an established diagnosis of IBD (Crohn's desease, ulcerative colitis, unclassified IBD or chronic pouchitis) will be eligible for inclusion in a consultation to schedule surgery or colonoscopy for disease relapse (at diagnosis or prior to initiation of treatment), irrespective of treatment received
  Interventions: Other: Collection of biological samples

INTERVENTIONS:
Other: Collection of biological samples — Collection of blood samples and intestinal biopsies during a surgery or colonoscopy for disease relapse

SUMMARY:
The CELESTE cohort will be a three-center prospective cohort associated with the creation of a biobank including Inflammatory Bowel Diseases (IBD) patients with active disease

DETAILED DESCRIPTION:
The CELESTE cohort will be a prospective cohort of IBD patients followed up at Nantes University Hospital, Jules Verne Clinic (Nantes) and/or Confluent Private Hospital (Nantes). The multicentric nature of the cohort including a tertiary referral center and two secondary care centers is a major asset, enabling the enrolment of a broad spectrum of patients, from those naïve to any immunomodulatory treatment to those refractory to multiple biologic therapies.

It will be associated with a multi-omics biobank with the aim of identifying new cellular and molecular signatures of success of the therapeutic strategy at one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Patients with an established diagnosis of IBD: CD, UC, unclassified IBD or refractory chronic pouchitis;
* Patients with active disease requiring surgery or endoscopy, whether performed at diagnosis or prior to initiation of new therapy;
* Patients who have given written consent to participate in the study and to keep biological samples for research purposes

Exclusion Criteria:

* Patients refusing to participate in the cohort;
* Patients with chronic inflammatory bowel disease quiescent at inclusion;
* Patients with a contraindication to general anaesthesia;
* Vulnerable patients (under court protection, curators, guardians);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients who are immunomodulator-naive or refractory to one or more lines of immunosuppressive, biotherapy, or small molecule therapy
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who succeed in their therapeutic strategy | One year after inclusion
  Determine the proportion of patients who succeed in their therapeutic strategy at one year

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Nantes, Nantes
  - Clinique Jules Verne, Nantes
  - Hopital Privé du Confluent, Nantes